CLINICAL TRIAL: NCT06593249
Title: Presentation, Management and Outcome of Tick-borne Encephalitis in Patients Referred to Infectious Diseases or Neurology
Brief Title: Management of Tick-borne Encephalitis
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: TBE in ID or Neurology
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2020-03

CONDITIONS: Infectious Encephalitis
Keywords: tick-borne encephalitis; outcome; neuroimaging; lumbar puncture; clinical management
MeSH Terms: conditions — Infectious Encephalitis; Encephalitis, Tick-Borne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TBE in Infectious Diseases Department: patients with TBE referred to ID
  Interventions: Other: No Intervention: Observational Cohort
- TBE in Neurology Department: Patients with TBE in Neurology Department
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — no intervention, observational study

SUMMARY:
In this retrospective cohort study of patients with tick-borne encephalitis (TBE), potential differences in the clinical presentation at admission and diagnostic and therapeutic management of patients with TBE initially referred to infectious diseases or neurology departments were assessed. Associations between severity of acute illness and clinical outcome were also explored.

ELIGIBILITY:
Inclusion Criteria:

* microbiologically confirmed tick-borne meningoencephalitis

Exclusion Criteria:

* Exchanged between ID and neurology within the first 48 hours due to organizational constraints
* Transferred from another hospital
* Lumbar puncture not performed
* Not fulfilling study criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tick-borne encepalitis referred to Infectious diseases or Neurology departments of the University Medical Centre Ljubljana, Slovenia during the COVID-19 pandemic (from March 2020 to September 2022).
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
head imaging | at admission
  Number (%) of patients with head imaging performed before proceeding to lumbar puncture.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljublajana, Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided
On reasonable request.